CLINICAL TRIAL: NCT02855905
Title: Year-round Health Enhancing Exercise and Coronary Artery Disease: Randomized Controlled Study
Brief Title: Year-round Health Enhancing Exercise and Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Finnish Institute of Occupational Health (Other); University of Texas Southwestern Medical Center (Other); Maastricht University (Other); Finnish Defense Forces (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: University of oulu/CadColdEx
Record Dates: First submitted 2016-06-23; First posted 2016-08-04 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Coronary Artery Disease
Keywords: Exercise; Cold Temperature
MeSH Terms: conditions — Coronary Artery Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Coronary artery disease patients (Experimental): Coronary artery disease patients are exposed to brief cold exposure (-15 C for 30 min) mainly subjected to facial region during which their cardiovascular responses are registered. Exposure was repeated 4 times: rest and exercise in 22 C and rest and exercise in -15 C.
  Interventions: Other: Exercise/Rest and cold/neutral temperature

INTERVENTIONS:
Other: Exercise/Rest and cold/neutral temperature — Subjects were either exercising or resting in either cold or neutral environmental temperature

SUMMARY:
A cold season involves higher cardiovascular morbidity and mortality. Several epidemiologic studies have implicated that persons with a cardiac disease, such as coronary artery disease (CAD) may be at higher risk for these adverse health events, but the mechanisms are not well established. Because both exercise and cold exposure stimulates cardiac and circulatory functions it is important to study their interaction especially among people with CAD and whose myocardial oxygen supply and function are weakened. The study examines how recommended health-enhancing upper and lower body exercise and warm-up in combination with cold exposure affects cardiovascular functions of people with CAD.

The research includes randomized controlled experiments where the participants are 35-75 year old men with CAD (CCS I-II) and recruited from the Oulu University Hospital. Each participant undergoes four different trials in random order where the temperature (+22°C or -15°C) and the form of exercise (brisk walking at 5.5 km/h or upper body exercise at 30 W), and warm-up regime is varied. The used exercise, clothing and exposure resemble an ordinary wintertime exercise event. Novel techniques are used to broadly assess cardiovascular function before, during and in the recovery phase.

The obtained information is synthesized and translated to tailored year-round exercise instructions for people with CAD by the research team including experts from sports sciences, physiology, public and occupational health, clinical sciences and with complementary knowledge in physical activity, effective interventions and cardiovascular function. The study has broad national and international impact on the relatively passive aging population having CAD and residing and working in a cold climate. The produced information enables finding means to activate persons with CAD and where appropriate and safe year-round exercise may reduce or prevent adverse health effects. Health care personnel will have an improved possibility to prescribe physical activity programs for their clients and enabling better instructions of healthy and safe exercise as a way to promote health.

DETAILED DESCRIPTION:
Introduction

National and International significance of the research

According to a worldwide estimate 42% of people with coronary artery disease (CAD) are physically inactive. There are approximately 200 000 persons in Finland with CAD, and even more have other connected health problems (high cholesterol or blood pressure, diabetes) further weakening their cardiac function and physical capacity and causing mortality. This increasing ageing population are often inactive, but would benefit substantially from regular year-round physical activity for maintaining their functional ability and independent living.

At present it is not known whether the exercise recommendation for CAD patients involves a health risk during cold exposure as they regularly report symptoms of chest pain and arrhythmias in the winter. Because both exercise and cold exposure stimulates cardiac and circulatory functions precise physical activity require defining their interaction among CAD patients whose myocardial oxygen supply and function are weakened.

Nationally and internationally the research addresses a large and special population group living in the northern hemisphere, whose symptoms, health events and mortality are common and provoked in the cold season. A passive lifestyle of this population is partially due to inadequate instructions and guidance. As a result of ageing the proportion of people with CAD will increase which emphasizes the role of prevention in reducing health care costs. The proposed research entity forms an important part of the research program examining the direct effect of temperature on human health in the newly established WHO Collaboration Centre in Global change, Environment and Public Health.

Aims and hypotheses The aims are: 1) to study separate and combined effects of upper or lower body exercise and warm-up on cardiovascular response (acute, recovery) and to 2) translate the research information into tailored instructions for year-round physical activity.

The hypotheses are: 1) moderate level endurance exercise increase cardiovascular strain in CAD patients in the cold compared to a warm environment, 2) upper body exercise is more strenuous than lower body exercise in the cold, 3) warm-up exercise attenuates the cold and exercise induced rise in BP

Participants The participants are 35-75-year old men (non-smokers) with CAD (NYHA CCS I-II), have experienced a myocardial infarction over 3 months ago, have hypertension but no other metabolic, cardiovascular or respiratory disease. The participants are recruited from the Oulu University Hospital by an experienced cardiologist. The exclusion criteria are: smoking, asthma, CCS class III-IV, diabetes, previous myocardial infarction less than 3 months ago, chronic atrial fibrillation, claudication, unstable angina pectoris, serious complex arrhythmias or ECG anomalies during rest.

Randomized controlled studies (n=160) The randomized controlled studies allow understanding causality and the physiological mechanisms for the separate and combined effects of exercise and cold on cardiovascular function in persons with CAD. Phase I (2015-16): Separate and combined effects of cold and exercise on cardiovascular function. Each participant (n=20) is randomly exposed to four conditions and separately to a neutral (+22°C) and cold (-15°C) environment during rest and exercise. Phase II (2016-17): Type of exercise and warm-up on cardiovascular function during exercise in the cold. Each participant (n=20) is randomly exposed to four conditions involving lower (brisk walking) or upper body (arm ergometry) exercise in the cold (-15°C) with or without warm-up exercise at +22°C. Each experimental session lasts for 105 min (15 min baseline + 30 min exposure + 60 min recovery).

Ambient conditions The participants are exposed to both +22°C and -15°C (wind 1.4. m/s) for 30 min per experimental session in the wind tunnel of the Kastelli Research Centre. The used cold exposure simulates conditions which occur frequently during the winter in a cold climate. The participants are equipped with winter clothing during the experiments. The cold exposure is largely restricted to the face which is known to increase BP by ca. 20 mmHg in healthy subjects.

Study protocol

The experimental sessions are performed at the same time of the day for each participant. Instructions to avoid heavy exercise or alcohol 48 h before or coffee/caffeine related beverages 3 h prior to the experiments are given. The participants are informed of the research, provide written consent to participate to the study and have a possibility to get acquainted with the experimental conditions. A questionnaire inquiring of the health and lifestyle of the participants is filled in. Following this the body composition of the subjects is assessed by bioimpedance. A baseline blood sample is drawn. After this the subjects are equipped with skin temperature thermistors and arm cuff (BP). ECG-electrodes are attached both for online (12-lead) and long term (24 h) monitoring of cardiac function. Subjects are followed in neutral conditions for 15 minutes (baseline). Continuous beat-to-beat BP, central aortic blood pressure and flow mediated dilation is recorded before the exposure to neutral/cold temperature and rest/exercise. For exercise in the cold the subjects are equipped with winter clothing and enter the experimental conditions (wind tunnel). During the exercise cardiovascular functions are followed continuously through the real-time ECG. BP is measured every third minute at rest and during exercise. Physical strain is assessed at 1- minute and thermal sensations at 5-minute intervals. The termination criteria include an ST-depression of more than 2 mm, symptoms of angina, as well as a sudden considerable change in BP. The termination of an experiment is decided by the paramedic nurse monitoring and medical doctor supervising the experimental session. After ending the exercise the cardiovascular functions are followed for 30 minutes at 22°C. A blood sample is taken immediately after the exercise. Continuous and central BP is measured 3-8 minutes following the exercise (early recovery) and after 15-20 minutes (delayed recovery). The subjects return 48-hours after the experiment for providing a blood sample which enables to examine both immediate and delayed effects on hematological parameters (blood coagulation factors, inflammation markers, endothelin).

Research environment and researchers

The research is coordinated by the Center for Environmental and Respiratory Health Research (CERH) at the University of Oulu and with co-operation from the Research Unit of Internal Medicine, Center for Machine Vision and Signal Analysis and Finnish, Institute of Occupational Health and Finnish Defence Forces. International co-operation includes the University of Texas Southwestern Medical Center and University of Maastricht. The experiments are conducted in the unique thermal laboratories of Kastelli Research Centre in Oulu with comprehensive and novel equipment for assessment of circulatory, respiratory, autonomic nervous system function and thermal balance. The research team is multidisciplinary and consists of experts of sports sciences, physiology, medicine, rehabilitation, and wellness technology.

Adjunct professor Tiina Ikäheimo (former Mäkinen), Ph.D., lecturer CERH, University of Oulu; PI of the research and with special expertise in physiology and the effects of temperature on human health and performance. The PI has produced several original publications and reviews and produced texts to national and international professional books (e.g. for WHO) of cold-related health risks and recommendations for their prevention.

Research group:

Professor Heikki Huikuri, MD, Ph.D., University of Oulu and Oulu University Hospital, Research Unit of Internal Medicine, Leader of Medical Research Center and expert in Cardiology; Adjunct professor Antti Kiviniemi, Ph.D., senior scientist of Exercise and Medical Physiology; Medical specialist in Cardiology, Juha Perkiömäki, MD, Ph.D.; Adjunct professor Mikko Tulppo, Ph.D.; Adjunct professor Arto Hautala, Ph.D. Center for Machine Vision and Signal Analysis, University of Oulu; Professor Markku Alén, MD, Ph.D., University of Oulu, Center for Life-Course Epidemiology (CLCE); Professor Hannu Rintamäki, Ph.D. Finnish Institute of Occupational Health; Professor Matti Mäntysaari*, MD, Ph.D., Director, Aeromedical Centre, Finnish Defence Forces; Professor Jouni J.K. Jaakkola, MD, Ph.D., Director, CERH, University of Oulu; Postgraduate student Heidi Hintsala, Master in Health Sciences (MHSc). CERH, University of Oulu; Professor emeritus Juhani Hassi, Ph.D. CERH, University of Oulu; Doctoral student Rasmus Valtonen, CERH University of Oulu; Paramedic nurse Miia Länsititie, CERH, University of Oulu, Project secretary Riitta Aittamaa, CERH, University of Oulu. INTERNATIONAL: Professor Craig Crandall, Ph.D., Division of Cardiology, Department of Internal Medicine, The University of Texas Southwestern Medical Center, USA. Professor Wouter van Marken Lichtenbelt, Ph.D. Health, Medicine and Life Sciences, Human Biology, Maastricht University, Netherlands.

Ethical questions

The study follows the declaration of Helsinki and the legislation, decrees and ethical principles concerning medical research on humans in Finland. The study has been approved by the Northern Ostrobothnia Hospital Districts Ethical Committee. The experimental tests are performed under the monitoring of a paramedic nurse and supervision of a medical doctor.

ELIGIBILITY:
Inclusion Criteria:

* CCS class I-II
* Non-smokers
* Hypertension
* Myocardial infarction over 3 months ago

Exclusion Criteria:

* smoking
* Asthma
* NYHA CCS class III-IV
* Diabetes
* Myocardial infarction less than 3 months ago
* Chronic atrial fibrillation
* Claudication
* Unstable angina pectoris
* Serious complex arrhythmias or ECG anomalies during rest.
* Bypass surgery
* Angioplasty

Ages: 35 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Blood pressure [mmHg, millimeter of mercury] | 3 hours
  Brachial blood pressure

SECONDARY OUTCOMES:
Electrocardiogram [mV, milliVolts] | 3 hours
  online 12-lead monitoring and data collection of cardiac electric activity
Flow-mediated dilation [arterial diameter mm, millimeter] | 3 hours
  ultrasound measurement of brachial blood flow following occlusion
Stress hormones (catecholamines) [nmol/l, nanomol / liter] | 3 hours
  collection of blood samples from where the following parameters are analysed: noradrenaline and adrenaline.
inflammatory markers [ng/l, nanogram / liter] | 3 hours
  collection of blood samples from where the following parameters are analysed: interleukin-6, c-reactive protein and (tumor necrosis factor) TNF-alpha
blood coagulation factors [mg/l, milligram / liter] | 3 hours
  collection of blood samples from where the following parameters are analysed: fibrinogen and protrombin
Skin temperature [°C, celsius] | 3 hours
  Skin temperature is measured by 8-channel temperature data loggers (SmartReaderPlus; Acr Systems, Surrey, BC, Canada). We have two data loggers and we use totally 10-channels. Thermistors are placed on the skin following places: right scapula, left side of the face, forehead, left calf, right anterior thigh, left index finger, left hand, left forearm, right shoulder, left upper chest.
Central aortic blood pressure [mmHg, millimeter of mercury] | 3 hours
  Central aortic BP is measured with the use of radial artery applanation tonometry. The measuring sensor is tonometric pressure sensor (SPC-301; Millar Instruments, Houston, Texas, USA). Tonometric pressure sensor is placed on the skin over the radial artery and the sensor transmits digitally the pulse of the artery.

CONTACTS AND LOCATIONS:
Overall Officials: Tiina M Ikäheimo, Ph.D., Principal Investigator — University of Oulu, Center for Environmental and Respiratory Health Research
Locations (1):
- University of Oulu, Center for Environmental and Respiratory Health Research, Oulu, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ikaheimo TM, Lehtinen T, Antikainen R, Jokelainen J, Nayha S, Hassi J, Keinanen-Kiukaanniemi S, Laatikainen T, Jousilahti P, Jaakkola JJ. Cold-related cardiorespiratory symptoms among subjects with and without hypertension: the National FINRISK Study 2002. Eur J Public Health. 2014 Apr;24(2):237-43. doi: 10.1093/eurpub/ckt078. Epub 2013 Jun 22. PMID 23794677
- [Result] Sun Z. Cardiovascular responses to cold exposure. Front Biosci (Elite Ed). 2010 Jan 1;2(2):495-503. doi: 10.2741/e108. PMID 20036896
- [Result] Hintsala H, Kandelberg A, Herzig KH, Rintamaki H, Mantysaari M, Rantala A, Antikainen R, Keinanen-Kiukaanniemi S, Jaakkola JJ, Ikaheimo TM. Central aortic blood pressure of hypertensive men during short-term cold exposure. Am J Hypertens. 2014 May;27(5):656-64. doi: 10.1093/ajh/hpt136. Epub 2013 Aug 20. PMID 23964061
- [Result] Hintsala H, Kentta TV, Tulppo M, Kiviniemi A, Huikuri HV, Mantysaari M, Keinanen-Kiukaannemi S, Bloigu R, Herzig KH, Antikainen R, Rintamaki H, Jaakkola JJ, Ikaheimo TM. Cardiac repolarization and autonomic regulation during short-term cold exposure in hypertensive men: an experimental study. PLoS One. 2014 Jul 1;9(7):e99973. doi: 10.1371/journal.pone.0099973. eCollection 2014. PMID 24983379
- [Result] Manou-Stathopoulou V, Goodwin CD, Patterson T, Redwood SR, Marber MS, Williams RP. The effects of cold and exercise on the cardiovascular system. Heart. 2015 May 15;101(10):808-20. doi: 10.1136/heartjnl-2014-306276. Epub 2015 Feb 11. No abstract available. PMID 25673528
- [Derived] Pikkarainen K, Valtonen RIP, Hintsala HE, Kiviniemi A, Crandall CG, Perkiomaki J, Hautala AJ, Tulppo MP, Jaakkola JJK, Ikaheimo TM. Baroreflex sensitivity following acute upper-body exercise in the cold among stable coronary artery disease patients. Front Physiol. 2023 Oct 13;14:1184378. doi: 10.3389/fphys.2023.1184378. eCollection 2023. PMID 37900953
- [Derived] Valtonen RIP, Hintsala HHE, Kiviniemi A, Kentta T, Crandall C, van Marken Lichtenbelt W, Perkiomaki J, Hautala A, Jaakkola JJK, Ikaheimo TM. Cardiovascular responses to dynamic and static upper-body exercise in a cold environment in coronary artery disease patients. Eur J Appl Physiol. 2022 Jan;122(1):223-232. doi: 10.1007/s00421-021-04826-x. Epub 2021 Oct 16. PMID 34655331
- [Derived] Hintsala HE, Valtonen RIP, Kiviniemi A, Crandall C, Perkiomaki J, Hautala A, Mantysaari M, Alen M, Ryti N, Jaakkola JJK, Ikaheimo TM. Central aortic hemodynamics following acute lower and upper-body exercise in a cold environment among patients with coronary artery disease. Sci Rep. 2021 Jan 28;11(1):2550. doi: 10.1038/s41598-021-82155-x. PMID 33510373
- [Derived] Ikaheimo TM, Lansitie M, Valtonen R, Hintsala HE, Ryti N, Perkiomaki J, Mantysaari M, Hautala AJ, Jaakkola JJK. Good safety practice in a randomized controlled trial (CadColdEx) involving increased cardiac workload in patients with coronary artery disease. BMC Cardiovasc Disord. 2019 Mar 25;19(1):69. doi: 10.1186/s12872-019-1051-1. PMID 30909877